CLINICAL TRIAL: NCT03114163
Title: A National, Prospective, Non-Interventional Study (NIS) of Nivolumab (BMS-936558) in Patients With Squamous Cell Carcinoma of the Head and Neck (SCCHN) Progressing on or After Platinum-Based Therapy
Brief Title: Observational Study of Nivolumab in Participants in Germany With Squamous Cell Carcinoma of the Head and Neck (SCCHN) Progressing on or After Platinum-Based Therapy
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: CA209-99K
Record Dates: First submitted 2017-04-10; First posted 2017-04-14 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Cohort 1: Nivolumab: ≥2nd line treatment for recurrent/ metastatic (R/M) Squamous cell carcinoma of the head and neck (SCCHN), prior platinum-based therapy was administered for locally advanced, metastatic or recurrent disease
- Cohort 2: Nivolumab: 1st line treatment for R/M SCCHN, prior platinum-based therapy was administered for locally advanced disease in the adjuvant or primary setting

SUMMARY:
This is a German, observational study in adult participants diagnosed with squamous cell carcinoma of the head and neck (SCCHN) progressing on or after platinum-based therapy, who start a new systemic therapy with nivolumab in 1st line (cohort 2) or ≥2nd line (cohort 1) for the first time, and are treated within the market authorization approval. Participants are to be enrolled into the study no earlier than the decision to initiate treatment with nivolumab and no later than the first dose of nivolumab treatment.

ELIGIBILITY:
For more information regarding Bristol-Myers Squibb Clinical Trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

- Adult participants (at least 18 years of age at time of treatment decision)

* Diagnosis of Squamous cell carcinoma of the head and neck (SCCHN) and participants are progressing on or after platinum-based therapy, administered for locally advanced, metastatic or recurrent disease (Cohort 2: prior platinum-based therapy was administered for locally advanced disease in the adjuvant or primary setting, e.g. radiotherapy)
* Diagnosis of SCCHN has been confirmed by histology or cytology (either at initial diagnosis or any time later during the course of the disease)
* Treatment decision to initiate a treatment with nivolumab for the first time for the treatment of SCCHN (according to the label approved in Germany) has already been taken

Exclusion Criteria:

* Current primary diagnosis of a cancer other than SCCHN, ie, a cancer other than SCCHN or cancer of unknown primary (CUP-syndrome) that requires systemic or other treatment, or has not been treated curatively (as per discretion of the investigator)
* Previously treated with nivolumab and/or ipilimumab, an anti-PD-1, anti-programmed death ligand 1 (anti-PD-L1), anti-PD-L2, anti-CTLA-4 antibody, or any other antibody or drug specifically targeting T-cell co-stimulation or immune checkpoint pathways (applicable for any indication)
* Currently included in an interventional clinical trial for their SCCHN. Participants who have completed their participation in an interventional trial; or who are not receiving study drug anymore and who are only followed-up for Overall survival (OS) can be enrolled

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will enroll adult participants who are at least 18 years of age at the time of the treatment decision, with the diagnosis of Squamous Cell Carcinoma of the Head and Neck (SCCHN) (either initial diagnosis or during later course histologically or cytologically confirmed). It is mandatory that the physician has already decided to initiate a treatment with nivolumab as 1st line or ≥2nd line therapy for the first time for the treatment of SCCHN, according to the label approved in Germany.
Sampling Method: Non-Probability Sample
Enrollment: 485 (Actual)
Dates: Start 2017-05-12 (Actual); Primary Completion 2025-04-28 (Actual); Study Completion 2025-04-28 (Actual)

PRIMARY OUTCOMES:
Overall Survival | Up to 5 years

SECONDARY OUTCOMES:
Overall Survival | Up to 5 years
Progression-Free Survival (PFS) | Up to 5 years
Time to progression | Up to 5 years
Overall Response Rate (ORR) | Up to 5 years
Best overall response rate (BORR) | Up to 5 years
Best overall response (BOR) | Up to 5 years
Tumor response (Investigator assessed) | Up to 5 years
Time to response (TTR) | Up to 5 years
Duration of response (DOR) | Up to 5 years
Description of socio-demographic characteristics of participants | Up to 5 years
Description of clinical characteristics of participants | Up to 5 years
Description of management of participants with treatment-related adverse events (AEs) | Up to 5 years
Description of incidence of AEs | Up to 5 years
Description of Severity of AEs | Up to 5 years
Description of management of AEs | Up to 5 years
Description of participant-reported outcomes (PROs) and health-related quality-of-life (QoL) of participants using the Functional Assessment of Cancer Therapy - Head & Neck (FACT-H&N) questionnaires | Up to 5 years
Description of participant-reported outcomes (PROs) and health-related quality-of-life (QoL) of participants using European Quality of Life-5 Dimensions (EQ-5D) questionnaires | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution - 0001, Leipzig, Germany

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/investigator-inquiry-form.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm